CLINICAL TRIAL: NCT03021824
Title: Severe ARDS: Generating Evidence. A U.S. Multicenter Observational Study.
Brief Title: Severe ARDS: Generating Evidence
Acronym: SAGE
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: University of Michigan (Other); Duke University (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-6757
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2019-12

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Respiratory Failure With Hypoxia; Acute Respiratory Failure
Keywords: Acute Respiratory Distress Syndrome; ARDS; Acute Lung Injury; ALI; Mechanical Ventilation; Extracorporeal Membrane Oxygenation; Neuromuscular Blockade; Vasodilator Agents; Prone Position; ECMO; Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Moderate-Severe ARDS: All adults admitted to participating ICUs with study-defined moderate-to-severe ARDS.

SUMMARY:
An assessment of early management of moderate-severe ARDS in the United States, including ventilator management and use of rescue therapy.

DETAILED DESCRIPTION:
Approximately one-quarter of ARDS patients develop severe hypoxemia, which has been associated with mortality rates approximating 40-50%. The majority have been described to present with severe disease at baseline, suggesting an opportunity for early intervention. In addition, use of evidence-based practices in severe ARDS is highly variable and inconsistent; use of unproven treatment modalities is also frequently seen. Given the variability in treatment practices in severe ARDS, an understanding of the patient-level and institutional-level factors contributing to differences in therapeutic approach is needed in order to improve the quality and consistency of care given to these high-risk patients. SAGE is a multicenter, observational cohort study examining the patient-level and institutional characteristics associated with variability in management of patients with moderate to severe ARDS, factors associated with survival or need for adjuvant therapy, and variability in ventilator management of patients on extracorporeal membrane oxygenation. Findings from this observational study can subsequently be used to inform future interventional trial development.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Patients with acute respiratory failure requiring invasive mechanical ventilation via an endotracheal tube or tracheostomy with current or planned admission to the ICU
3. Moderate-severe ARDS as defined by fulfillment of all of the following within 48 hours:

   1. Bilateral opacities detected on chest radiograph or CT, not fully explained by effusions, lung collapse, or nodules
   2. Respiratory failure not fully explained by cardiac failure or fluid overload
   3. PaO2/FiO2 ratio < 150 with a minimum of 5 cmH20 PEEP

Exclusion Criteria:

There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults admitted to participating ICUs with study-defined moderate-to-severe ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | 28 Days
Use of Adjunctive Therapy | 28 Days

SECONDARY OUTCOMES:
Ventilator-Free Days | 28 Days
ICU-Free Days | 28 Days
Organ Failure | 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Nida Qadir, MD, Principal Investigator — Montefiore Medical Center; Pauline Park, MD, Principal Investigator — University of Michigan; Raquel Bartz, MD, Principal Investigator — Duke University; Michelle N Gong, MD, Principal Investigator — Montefiore Medical Center
Locations (28):
- United States (28):
  - University of Arizona, Tucson, Arizona
  - Los Angeles County + University of Southern California Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Saint Joseph Mercy Ann Arbor, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Northwell Health, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregan Health and Science University Hospital, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Qadir N, Bartz RR, Cooter ML, Hough CL, Lanspa MJ, Banner-Goodspeed VM, Chen JT, Giovanni S, Gomaa D, Sjoding MW, Hajizadeh N, Komisarow J, Duggal A, Khanna AK, Kashyap R, Khan A, Chang SY, Tonna JE, Anderson HL 3rd, Liebler JM, Mosier JM, Morris PE, Genthon A, Louh IK, Tidswell M, Stephens RS, Esper AM, Dries DJ, Martinez A, Schreyer KE, Bender W, Tiwari A, Guru PK, Hanna S, Gong MN, Park PK; Severe ARDS: Generating Evidence (SAGE) Study Investigators; Society of Critical Care Medicine's Discovery Network. Variation in Early Management Practices in Moderate-to-Severe ARDS in the United States: The Severe ARDS: Generating Evidence Study. Chest. 2021 Oct;160(4):1304-1315. doi: 10.1016/j.chest.2021.05.047. Epub 2021 Jun 4. PMID 34089739